CLINICAL TRIAL: NCT01147237
Title: A Multi Center Registry to Evaluate Multiple Stenting Using by Everolimus-eluting Stents for Treatment of Long Coronary Artery Disease
Brief Title: Xience/Promus for Long Coronary Lesion Registry
Acronym: XILLION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Society for Advancement of Coronary Intervention Research (Network)
Responsible Party: Kenya Nasu, Toyohashi Heart Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XILLION
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Long Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Experimental)
  Interventions: Device: Intracoronary stent implantation

INTERVENTIONS:
Device: Intracoronary stent implantation — Everolimus-eluting stent implantation in patients with long coronary artery disease

SUMMARY:
The utilization of everolimus-eluting coronary stents in a coronary artery diseases is effective in reducing both repeat revascularization and major adverse cardiac events within two year follow-up. To evaluate the procedural, short and long term clinical outcomes of multiple everolimus-eluting coronary stent implantation in long (>30mm) coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 years and are able to undergo CABG
2. Females who are not pregnant
3. Patients who present with angina symptoms or myocardial ischemia
4. Patients available for post-procedural observation and coronary angiography at 24 months
5. Patients who have signed patient informed consent
6. Lesion length is more than 30mm
7. De novo lesion or non-stented restenosed lesion

Exclusion Criteria:

1. Patients contraindicated for antiplatelet therapy or anticoagulant therapy
2. Patients with significant allergic reaction to contrast medium
3. Chronic total occlusion
4. Lesion with TIMI0
5. Patients with chronic renal failure (SCr>3.0mg/dl) -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Target lesion revascularization rate | 1 year

SECONDARY OUTCOMES:
Technical success | Initial
Angiographic restenosis | 9 months
Target vessel revascularization | 1 year
Target lesion revascularization | 2 year
Target vessel revascularization | 2 year
Incidences of acute, sub acute, and late stent thrombosis | 2 year
Incidence of MACCE | 2 year
  defined as cardiac death, nonfatal acute myocardial infarction and cerebrovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Oikawa, MD, PhD, Principal Investigator — Cardiovascular institute hospital; Kenya Nasu, MD, Principal Investigator — Toyohashi Heart Center
Locations (31):
- Japan (31):
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - Toyohashi Heart Center, Toyohashi, Aichi-ken
  - Higashi Cardiovascular clinic, Toyohashi, Aichi-ken
  - Hiraka General Hospital, Yokote, Akita
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - Kokura memorial hospital, Kitakyushu, Fukuoka
  - Hoshi General Hospital, Kōriyama, Fukushima
  - Gunma Prefectural Cardiovascular Center, Maebashi, Gunma
  - Abashiri Kosei General Hospital, Abashiri, Hokkaido
  - Engaru-Kosei General Hospital, Engaru, Hokkaido
  - Hakodate Goryokaku Hospital, Hakodate, Hokkaido
  - Obihiro National Hospital, Obihiro, Hokkaido
  - Kinikyo Chuo Hospital, Sapporo, Hokkaido
  - Sapporo Orthopaedic Cardiovascular Hospital, Sapporo, Hokkaido
  - Shinko Kakogawa Hospital, Kakogawa, Hyōgo
  - Daini Okamoto Hospital, Uji, Kyoto
  - Miyagi Cardiovascular ＆ Respiratory Center, Kurihara, Miyagi
  - Matsumoto Kyoritsu Hospital, Matsumoto, Nagano
  - Rinku General Medical Center, Izumiōtsu, Osaka
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - Shuwa General Hospital, Kasukabe, Saitama
  - Kusatsu Heart Center, Kusatsu, Shiga
  - Ayase Heart Hospital, Adachi City, Tokyo
  - Juntendo University Hospital, Bunkyo, Tokyo
  - Tokyo-kita Social Insurance Hospital, Kita-ku, Tokyo
  - Cardiovascular Institute Hospital, Minato-ku, Tokyo
  - JR Tokyo General Hospital, Shibuya City, Tokyo
  - Tokyo Medical University Hospital, Shinjuku, Tokyo
  - Itabashi Chuo Medical Center, tabashi City, Tokyo
  - Tokyo Metropolitan Police Hospital, Tokyo, Tokyo